CLINICAL TRIAL: NCT02658669
Title: Cognitive Behavioral Therapy for Insomnia for Veterans With History of TBI
Brief Title: Cognitive-Behavioral Therapy for Veterans With TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D1512-W
Record Dates: First submitted 2016-01-11; First posted 2016-01-20 (Estimated); Results first posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-08

CONDITIONS: Insomnia; Traumatic Brain Injury
Keywords: Insomnia; Injury, Brain, Traumatic Mild
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Brain Injuries, Traumatic; Brain Concussion | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive-Behavioral Therapy for Insomnia (Experimental): 6-week manualized treatment designed to improve symptoms of chronic insomnia.
  Interventions: Behavioral: Cognitive-Behavioral Therapy for Insomnia
- Sleep Education (Active Comparator): 6-week manualized treatment designed to provide information regarding traumatic brain injury and its relationship to sleep disturbance, which incorporates training in sleep hygiene to help improve nighttime sleep and daytime functioning.
  Interventions: Behavioral: Sleep Education

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy for Insomnia — Intervention includes strategies designed to improve sleep such as: sleep restriction, stimulus-control techniques, sleep hygiene education, and relaxation training.
  Other Names: CBT-I
  Arms: Cognitive-Behavioral Therapy for Insomnia
Behavioral: Sleep Education — Intervention includes sleep hygiene education and education regarding the impact of TBI on sleep.
  Arms: Sleep Education

SUMMARY:
Many Operation Enduring Freedom/Operation Iraqi Freedom/Operation New Dawn era Veterans have suffered a mild traumatic brain injury (mTBI), and now cope with multiple post-injury symptoms, including sleep disturbances (especially insomnia). Chronic insomnia in mTBI patients has the potential to exacerbate other symptoms, delay recovery, and negatively affect many of the cognitive, psychological, and neuromuscular sequelae of mTBI, thereby decreasing quality of life. Although Cognitive-Behavioral Therapy for Insomnia (CBT-I) has been shown to be an effective evidence-based treatment for insomnia, there are no published randomized controlled trials evaluating the potential strengths and/or limitations of CBT-I in post-mTBI patients. Therefore, assessing CBT-I in the context of mTBI holds promise to provide substantial benefits in terms of improved rehabilitation outcomes in Veterans who have suffered mTBI.

DETAILED DESCRIPTION:
This VA Rehabilitation Research and Development Career Development Award (CDA-2) proposal is designed to significantly advance the application of Behavioral Sleep Medicine practices in the treatment of Veterans seen in the VA Healthcare System, especially those recovering from traumatic brain injury (TBI). TBI has been deemed the "signature wound" of the Iraq and Afghanistan Wars, occurring in about 19.5% of Operation Enduring Freedom/Operation Iraqi Freedom/Operation New Dawn (OEF/OIF/OND) service members. For many Veterans, mild traumatic brain injury (mTBI) can be associated with persistent post-concussive symptoms, especially sleep disturbances. Sleep disturbances are among the most frequent complaints following mTBI, with studies suggesting that over 93% of Veterans who experienced brain injuries develop chronic sleep problems. Of the sleep disturbances diagnosed in this patient population the most common is insomnia, observed in over 50% of patients. Chronic and untreated insomnia is known to be associated with and/or increase risk for psychiatric problems, suicidal ideation, and unhealthy lifestyles (e.g., alcohol/drug abuse), lead to poorer physical health, disruption in major social and occupational responsibilities, and decreased quality of life, and may generally contribute to the persistence of post-concussive symptoms beyond the expected period of recovery. As such, treatment of sleep disturbance represents an essential component of Veteran care, one which may be particularly beneficial for Veterans with history of mTBI who commonly present to the clinic with complex multi-symptom concerns.

To address this important clinical issue, the proposed randomized clinical trial (RCT) will attempt to assess the efficacy of Cognitive-Behavioral Therapy for Insomnia (CBT-I) versus a Sleep Education control in Veterans with insomnia and a history of mTBI. CBT-I is recommended by the American Academy of Sleep Medicine for treatment of chronic insomnia and has also been adopted by the VA within an Evidence Based Practice roll-out program. Despite the acceptance of CBT-I as a first line treatment for sleep disturbance, there are no published RCTs evaluating CBT-I in mTBI patient populations. Therefore, this proposed investigation will address this gap in the literature by assessing the efficacy of CBT-I in Veterans with history of head injury.

ELIGIBILITY:
Inclusion Criteria:

1. OEF/OIF/OND Veteran ages 18-55.
2. Documented history of mild TBI (documented in the medical record and where possible from the VA TBI second-level evaluation)

   1. Loss of consciousness 30 minutes
   2. Post-traumatic amnesia 1 day
3. At least 3 months post-TBI.
4. A diagnosis of insomnia classified as:

   1. Diagnostic and Statistical Manual of Mental Disorders-5 (DSM 5) criteria that include: trouble falling asleep, staying asleep, waking too early, and/or non-restorative sleep with accompanied daytime impairment in functioning for > 3 months, occurring at least 3 nights per week.
   2. Subjective sleep disturbance defined by a Pittsburgh Sleep Quality Index score >5 and Insomnia Severity Index score >7 at intake.
5. No prior exposure to and/or treatment with CBT-I within the past 2 years.
6. Must be stable on medication regimen for at least 1 month prior to enrollment in study.

Exclusion Criteria:

1. History of a neurological disorder (besides TBI), dementia, or premorbid IQ <70.
2. Schizophrenia, psychotic disorder, and/or bipolar disorder.
3. Evidence of suicidality more than "low risk" as determined by the VA Comprehensive Suicide Risk Assessment (CSRA).
4. Sleep disturbances other than insomnia (e.g., untreated obstructive sleep apnea and/or periodic limb movements)
5. Alcohol and/or substance abuse within the past 30 days.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry J. Orff, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The SRS fosters scientific investigations on all aspects of sleep and its disorders. — http://www.sleepresearchsociety.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Number of participants enrolled (73) differs from participants started due to lack of eligibility post consent/baseline or declining continued participation.
Period: Overall Study
Arm/Group | Cognitive-Behavioral Therapy for Insomnia | Sleep Education
Started | 27 | 28
Completed | 20 | 23
Not Completed | 7 | 5
Not completed — Lost to Follow-up | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive-Behavioral Therapy for Insomnia | Sleep Education | Total
Number analyzed (Participants) | 27 | 28 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (6.7) | 34.75 (7.1) | 36.0 (6.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 20 | 25 | 45
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Insomnia Severity
Description: Change in insomnia severity. Scale used is Insomnia Severity Index (ISI). Minimum value= 0; maximum value = 28. Lower score equals better outcome.
Time Frame: Pre-Treatment (0-weeks), Post-Treatment (8-weeks), Follow-Up (12-weeks)
Population: Overall number of participants analyzed reflects patients assessed at week 0, and total number analyzed reflected patients who were assessed at later time points. Differences due to drop-out of patients in the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive-Behavioral Therapy for Insomnia | Sleep Education
Number analyzed (Participants) | 26 | 28
score on a scale
  ISI Pre to Post: number analyzed (Participants) | 18 | 21
  ISI Pre to Post | 8.833 (4.743) | 7.810 (7.366)
  ISI Pre to Follow-Up: number analyzed (Participants) | 8 | 11
  ISI Pre to Follow-Up | 9.625 (5.927) | 8.364 (8.250)

2. Secondary Outcome: Change in Depressive Symptomatology
Description: Change in depressive symptoms assessed using the Patient Health Questionnaire-9 (PHQ-9) a self-report measure of depression. Minimum value = 0; maximum value = 27. Lower scores indicate fewer depressive symptoms.
Time Frame: Pre-Treatment (0-weeks), Post-Treatment (8-weeks), Follow-Up (12-weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive-Behavioral Therapy for Insomnia | Sleep Education
Number analyzed (Participants) | 26 | 28
score on a scale
  PHQ-9 Pre to Post: number analyzed (Participants) | 19 | 23
  PHQ-9 Pre to Post | 3.789 (5.534) | 1.609 (4.659)
  PHQ-9 Pre to Follow-Up: number analyzed (Participants) | 8 | 12
  PHQ-9 Pre to Follow-Up | 3.250 (5.312) | -2.250 (16.907)

3. Secondary Outcome: Change in PTSD Stressor Specific Checklist 5
Description: Change in PTSD symptoms assessed using the PTSD Stressor Specific Checklist 5 (PCL-5) a self-report measure of PTSD. Minimum score = 0, maximum score = 80. Lower scores indicate less PTSD symptomatology.
Time Frame: Pre- Treatment (0-weeks), Post-Treatment (8-weeks), Follow-Up (12-weeks)
Population: Difference in overall number of participants and number analyzed differs due to lack of completion of treatment. Overall number refers to those who were assessed at week-0 treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive-Behavioral Therapy for Insomnia | Sleep Education
Number analyzed (Participants) | 26 | 28
score on a scale
  PCL-5 Pre to Post: number analyzed (Participants) | 19 | 22
  PCL-5 Pre to Post | 8.053 (13.373) | 6.227 (10.497)
  PCL-5 Pre to Follow-Up: number analyzed (Participants) | 8 | 11
  PCL-5 Pre to Follow-Up | 3.125 (12.822) | 4.727 (11.516)

4. Secondary Outcome: Change in World Health Organization Disability Assessment Scale-2
Description: Change in global functioning and disability will be assessed using the World Health Organization Disability Assessment Scale-2, a self-report measure. Minimum value = 0; maximum value = 100. Lower scores indicates less disability.
Time Frame: Pre- Treatment (0-weeks), Post-Treatment (8-weeks), Follow-Up (12-weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive-Behavioral Therapy for Insomnia | Sleep Education
Number analyzed (Participants) | 26 | 28
score on a scale
  WHODAS Pre to Post: number analyzed (Participants) | 19 | 22
  WHODAS Pre to Post | -0.316 (25.478) | 1.818 (14.702)
  WHODAS Pre to Follow-Up: number analyzed (Participants) | 5 | 11
  WHODAS Pre to Follow-Up | 17.200 (18.754) | 8.273 (19.032)

5. Secondary Outcome: Change in Pittsburgh Sleep Quality Index
Description: Change in sleep quality will be assessed with the Pittsburgh Sleep Quality Index (PSQI). Minimum value = 0; maximum value= 21. Lower score indicates less general sleep disturbance.
Time Frame: Pre- Treatment (0-weeks), Post-Treatment (8-weeks), Follow-Up (12-weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive-Behavioral Therapy for Insomnia | Sleep Education
Number analyzed (Participants) | 26 | 28
score on a scale
  PSQI Pre to Post: number analyzed (Participants) | 17 | 20
  PSQI Pre to Post | 5.412 (3.183) | 4.400 (3.633)
  PSQI Pre to Follow-Up: number analyzed (Participants) | 8 | 12
  PSQI Pre to Follow-Up | 5.125 (2.748) | 4.833 (4.821)

6. Other Pre Specified Outcome: Change in Patient Reported Outcomes Measurement Information System (PROMIS) Pain
Description: Change in pain will be assessed using the Patient Reported Outcomes Measurement Information System (PROMIS) pain assessment, as self-report measure of pain. Measures are scored on a T-score (mean=50, SD=10) Minimum score = <20 ; maximum score = >80. Lower scores indicate less pain interference in daily life.
Time Frame: Pre- Treatment (0-weeks), Post-Treatment (8-weeks), Follow-Up (12-weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive-Behavioral Therapy for Insomnia | Sleep Education
Number analyzed (Participants) | 26 | 28
score on a scale
  PROMIS Pre to Post: number analyzed (Participants) | 15 | 18
  PROMIS Pre to Post | -0.8333 (4.4042) | 3.3778 (5.4668)
  PROMIS Pre to Follow-Up: number analyzed (Participants) | 7 | 12
  PROMIS Pre to Follow-Up | -2.5714 (5.1768) | 2.050 (2.1581)

7. Other Pre Specified Outcome: Change in Neuropsychological Functioning: Attention/Processing Speed
Description: Change in cognitive functioning will be evaluated through standardized assessments of attention and processing speed. The tasks that will be administered include: the Wechsler Adult Intelligence Scale Fourth Edition (WAIS-IV) Digit Symbol and Symbol Search to measure attention and processing speed. WAIS-IV raw minimum value score=45; maximum score=155. Scaled score used: minimum score = 1; maximum score = 19. Higher score equals a better outcome.
Time Frame: Pre- Treatment (0-weeks), Post-Treatment (8-weeks), Follow-Up (12-weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive-Behavioral Therapy for Insomnia | Sleep Education
Number analyzed (Participants) | 26 | 28
score on a scale
  Symbol Search WAIS Pre to Post: number analyzed (Participants) | 10 | 17
  Symbol Search WAIS Pre to Post | -1.90 (3.035) | -0.882 (2.395)
  Symbol Search WAIS Pre to Follow-Up: number analyzed (Participants) | 5 | 10
  Symbol Search WAIS Pre to Follow-Up | -3.400 (2.302) | -1.200 (3.765)
  Coding WAIS Pre to Post: number analyzed (Participants) | 9 | 18
  Coding WAIS Pre to Post | -0.667 (1.000) | -1.500 (2.875)
  Coding WAIS Pre to Follow-Up: number analyzed (Participants) | 5 | 10
  Coding WAIS Pre to Follow-Up | -2.600 (2.608) | -1.100 (3.784)

8. Other Pre Specified Outcome: Change In Neuropsychological Functioning: Verbal Learning and Memory
Description: Change in cognitive functioning will be evaluated through standardized assessments of verbal learning and memory. The Hopkins Verbal Learning Test-Revised (HVLT-R) was used to measure learning and memory, and was measured by "Total Recall" score and "Delayed Recall" score. HVLT Total Recall raw scores minimum value=0; maximum value=36. Measures scored on a T-Score; minimum t-score score:0, maximum t-score >80. Higher t-scores indicate better outcome. HVLT delayed recall minimum raw score value=0; maximum value=12. Measures scored on a T-Score; maximum t-score value: 60, minimum =0. Higher t-scores indicate better outcome. Population mean and standard deviation calculated based on age. Mean age of the population was 36 years = total recall population t score mean: 28.04, SD: 4.43. Delayed recall population t score mean: 9.92, SD: 2.04.
Time Frame: Pre- Treatment (0-weeks), Post-Treatment (8-weeks), Follow-Up (12-weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive-Behavioral Therapy for Insomnia | Sleep Education
Number analyzed (Participants) | 26 | 28
score on a scale
  HVLT Total Pre to Post T-Score: number analyzed (Participants) | 9 | 20
  HVLT Total Pre to Post T-Score | -0.111 (8.937) | -1.099 (10.228)
  HVLT Total Pre to Follow-Up T-Score: number analyzed (Participants) | 5 | 10
  HVLT Total Pre to Follow-Up T-Score | -4.200 (10.426) | -8.200 (7.613)
  HVLT Delayed Pre to Post T-Score: number analyzed (Participants) | 9 | 20
  HVLT Delayed Pre to Post T-Score | -4.556 (7.485) | -7.300 (14.914)
  HVLT Delayed Pre to Follow-Up T-Score: number analyzed (Participants) | 5 | 10
  HVLT Delayed Pre to Follow-Up T-Score | -3.200 (9.985) | -12.000 (13.030)

9. Other Pre Specified Outcome: Change In Neuropsychological Functioning: Executive Functioning
Description: Change in cognitive functioning will be evaluated through standardized assessments of executive functioning. The Delis-Kaplan Executive Function Scale (D-KEFS) Trials and Color-Word Tasks was used to measure executive functioning, as measured by Color-Word Inhibition, Color-Word Switching Inhibition, and Trails. Scored using a scaled-score (minimum=1, maximum=19 for all measures). Higher scores indicate better outcome.
Time Frame: Pre- Treatment (0-weeks), Post-Treatment (8-weeks), Follow-Up (12-weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive-Behavioral Therapy for Insomnia | Sleep Education
Number analyzed (Participants) | 26 | 28
score on a scale
  DKEFS Color-Word Inhibition Pre to Post: number analyzed (Participants) | 9 | 20
  DKEFS Color-Word Inhibition Pre to Post | -1.333 (1.803) | -0.850 (2.412)
  DKEFS Color-Word Inhibition Pre to Follow-Up: number analyzed (Participants) | 5 | 10
  DKEFS Color-Word Inhibition Pre to Follow-Up | -1.400 (2.074) | -0.700 (1.494)
  DKEFS Color Word Inhibition Switching Pre to Post: number analyzed (Participants) | 9 | 20
  DKEFS Color Word Inhibition Switching Pre to Post | -1.667 (1.581) | -1.850 (2.059)
  DKEFS Color Word Inhibition Switching Pre to Follow-Up: number analyzed (Participants) | 5 | 10
  DKEFS Color Word Inhibition Switching Pre to Follow-Up | -1.00 (1.581) | -2.200 (2.530)
  DKEFS Trails Pre to Post: number analyzed (Participants) | 9 | 17
  DKEFS Trails Pre to Post | -0.667 (1.581) | -0.353 (1.169)
  DKEFS Trails Pre to Follow-Up: number analyzed (Participants) | 5 | 10
  DKEFS Trails Pre to Follow-Up | -1.400 (2.074) | -0.700 (1.418)

10. Other Pre Specified Outcome: Change in Sleep Efficiency as Measured by Polysomnography
Description: Change in sleep efficiency will be assessed through overnight polysomnographic sleep studies.
Time Frame: Pre-Treatment (0-weeks),Post-Treatment (8-weeks), Follow-Up (12-weeks)
Population: Data not collected due to pandemic.
Arm/Group | Cognitive-Behavioral Therapy for Insomnia | Sleep Education
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 12 weeks, through study completion and follow-up
Arm/Group | Cognitive-Behavioral Therapy for Insomnia | Sleep Education
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/28
Other Adverse Events (participants affected / at risk) | 0/27 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-26): https://cdn.clinicaltrials.gov/large-docs/69/NCT02658669/Prot_SAP_000.pdf